CLINICAL TRIAL: NCT00419419
Title: Phase III "In-Life" Study of a Topical Gel Formulation of Nitroglycerin, MQX-503, and Matching Placebo Gel in the Treatment and Prevention of Raynaud's Phenomenon
Brief Title: Phase III Study of a Topical Gel Formulation for Treatment and Prevention of Raynaud's Phenomenon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MediQuest Therapeutics (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 06-005
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Raynaud's Disease; Scleroderma; Autoimmune Diseases
Keywords: Raynaud's
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse; Autoimmune Diseases | interventions — Nitroglycerin

INTERVENTIONS:
Drug: Topical AmphiMatrix with nitroglycerin (MQX-503)

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of Topical AmphiMatrix with Nitroglycerin (MQX-503) to relieve Raynaud's symptoms and increase blood flow to the fingers.

DETAILED DESCRIPTION:
The purpose of this clinical study is to determine, in a controlled fashion, the ability of Topical AmphiMatrix formulation with Nitroglycerin (MQX-503) to improve the patient's health assessment as indicated by patient and physician assessments, decrease the frequency of Raynaud's events, decrease the duration of Raynaud's events, and decrease the symptoms (pain, tingling, numbness) in the fingers of Raynaud's patients. The study will include patients with moderate to severe primary Raynaud's phenomenon and with Raynaud's phenomenon secondary to autoimmune diseases such as scleroderma.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, 18 years to 70 years.
* Patients with a clinical diagnosis of Raynaud's phenomenon.
* Patients who are willing to discontinue current vasodilator therapies.
* Patients who agree not to use any other investigational medications or approved therapies to treat Raynaud's phenomenon and its symptoms while participating in this study.
* Negative pregnancy test in fertile women.
* Patients who are able to give written informed consent and comply with all study requirements.

Exclusion Criteria:

* Patients who concurrently use any nitrate medication or medications known to interact with Nitroglycerin.
* Patients who concurrently use any medication or device which might interfere with the study medication.
* Patients who have a known allergy to Nitroglycerin or common topical gel ingredients.
* Patients with a history of headaches.
* Patients who have a history of an unstable medical problem.
* Patients with cognitive or language difficulties.
* Patients who, within the past three months, have had either a myocardial infarction, uncontrolled congestive heart failure, unstable angina, uncontrolled hypotension, or uncontrolled hypertension.
* Patients who participated in a study of any investigational drug within four weeks prior to Visit 1.
* Patients who have screening laboratory values which are 20% or greater of the upper or lower limit of normal.
* Patients who have had major surgery within six months of Visit 1.
* Patients with interfering skin conditions.
* Pregnant or nursing women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-12

PRIMARY OUTCOMES:
Reduction in Raynaud's Condition Score

SECONDARY OUTCOMES:
Frequency and Severity of adverse events

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - Standford Medical School, Stanford, California
  - University of Connecticut, Farmington, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - The Center for Rheumatology, Albany, New York
  - Duke University, Durham, North Carolina
- Lund University Hospital, Lund, Sweden
- United Kingdom (5):
  - Royal National Hospital for Rheumatic Diseases, Bath
  - Ninewells Hospital and Medical School, Dundee
  - University of Leeds, Leeds
  - Royal Free Hospital, London
  - Hope Hospital, Salford